CLINICAL TRIAL: NCT05701449
Title: Prevention and Treatment of Perioperative Lung Injury in Elderly Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: China-Japan Friendship Hospital (Other); Taihe Hospital (Other); Chinese PLA General Hospital (Other); First Affiliated Hospital of Zhejiang University (Other); First Affiliated Hospital of Guangxi Medical University (Other); Qinghai People's Hospital (Other); Shanxi Cardiovascular Hospital (Other); Wuhan No.1 Hospital (Other); Shiyan City Renmin Hospital (Other Government); Dongfeng General Hospital of Chinese Medicine (Unknown); Xiangyang Central Hospital (Other); Xiangyang No.1 People's Hospital (Other); Hubei University of Medicine (Other); Yunxi Renmin Hospital (Unknown); Yunyang Renmin Hospital (Unknown); Zhuxi Renmin Hospital (Unknown); Danjiangkou First Hospital (Unknown); Shiyan Integrated Traditional and Western Medicine Hospital (Unknown); Shiyan Traditional Chinese Medicine Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: PPCS192023
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Postoperative Pulmonary Complications; Elderly Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients applying a prediction model for postoperative pulmonary complications
- Patients non-applying a prediction model for postoperative pulmonary complications

SUMMARY:
This study aims to verify the prediction model of postoperative pulmonary complications by collecting clinical information on elderly patients. In addition, the incidence of postoperative pulmonary complications in elderly patients before and after using the prediction model was compared.

DETAILED DESCRIPTION:
More than 300 million major operations are performed worldwide each year, and older patients account for about a third of elective operations. Compared with young people, the elderly are more prone to postoperative complications due to age-related degeneration of the physiological functions of various organs and tissues. Postoperative pulmonary complications, including pneumonia, atelectasis, and respiratory failure, are common. Even mild pulmonary complications can lead to the prolonged hospital stay and increased postoperative mortality.

Although there have been many studies on postoperative lung complications, there have been few studies on elderly patients. In our country, the real incidence data of elderly patients after a perioperative period of pulmonary complications, the lack of effective prevention, intervention measures, and targeted prevention and treatment technology, these reasons lead to the clinical diagnosis and treatment of elderly patients after a perioperative period of pulmonary complications are very difficult. Therefore, the research team intends to verify the established prediction model of postoperative pulmonary complications and compare the incidence of postoperative pulmonary complications in elderly patients before and after using the prediction model.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65 years or older
2. receiving invasive ventilation during general anesthesia for surgery

Exclusion Criteria:

1. preoperative mechanical ventilation
2. procedures related to a previous surgical complication
3. a second operation after surgery within one week
4. organ transplantation
5. discharged within 24 hours after surgery

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Patients aged 65 years or older
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative pulmonary complications | within one week after surgery

SECONDARY OUTCOMES:
Length of postoperative hospital stay | 6 weeks after surgery
Postoperative Death | 6 weeks after surgery